CLINICAL TRIAL: NCT01146392
Title: A Retrospective Epidemiological Study to Map Out Patients With Chronic Obstructive Pulmonary Disease (COPD) and Describe COPD Health Care in Real-Life Primary Care During the First Ten Years of the 21th Century
Brief Title: An Investigation of the Past 10 Yrs Health Care for Primary Care Patients With Chronic Obstructive Pulmonary Disease
Acronym: PATHOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RSE-DUM-2010/1
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Epidemiological; COPD health care; treatment in primary care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Primary care patients with COPD diagnosis

SUMMARY:
The aim of this study is to describe COPD health care and to assess demographics, concurrent diseases and mortality and the use of pharmaceuticals for a chronic obstructive pulmonary disease (COPD) population in real life in primary care during the last ten years.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to medical records.
* Use of drugs prescribed for obstructive lung diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects are all COPD patients, found in medical records at the participating swedish primary care clinics. Primarily patients with diagnosis code J44 (ICD-10) stated in the medical record will be investigated. Patient data from the period 1 January 1999 - 31 December 2009 will be included in the observation.
Sampling Method: Non-Probability Sample
Enrollment: 27394 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Describe the development of COPD health care structure in primary care. | Data will be extracted from the medical records on one occassion, covering a period of one decade.

SECONDARY OUTCOMES:
Describe the COPD population in primary care with special reference to treatment, co-morbidity and mortality during last decade. | Data will be extracted from the medical records on one occassion, covering a period of one decade.

CONTACTS AND LOCATIONS:
Overall Officials: Docent Gunnar Johansson, Principal Investigator — Uppsala University, Sweden; Kjell Larsson, Prof, Study Chair — Karolinska Institutet; Georgios Stratelis, MD, Study Director — AstraZeneca Nordics
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Result] Larsson K, Janson C, Lisspers K, Jorgensen L, Stratelis G, Telg G, Stallberg B, Johansson G. Combination of budesonide/formoterol more effective than fluticasone/salmeterol in preventing exacerbations in chronic obstructive pulmonary disease: the PATHOS study. J Intern Med. 2013 Jun;273(6):584-94. doi: 10.1111/joim.12067. Epub 2013 Apr 1. PMID 23495860
- [Result] Stallberg B, Janson C, Johansson G, Larsson K, Stratelis G, Telg G, Lisspers KH. Management, morbidity and mortality of COPD during an 11-year period: an observational retrospective epidemiological register study in Sweden (PATHOS). Prim Care Respir J. 2014 Mar;23(1):38-45. doi: 10.4104/pcrj.2013.00106. PMID 24346825
- [Derived] Sandelin M, Mindus S, Thuresson M, Lisspers K, Stallberg B, Johansson G, Larsson K, Janson C. Factors associated with lung cancer in COPD patients. Int J Chron Obstruct Pulmon Dis. 2018 Jun 6;13:1833-1839. doi: 10.2147/COPD.S162484. eCollection 2018. PMID 29922050
- [Derived] Lisspers K, Johansson G, Jansson C, Larsson K, Stratelis G, Hedegaard M, Stallberg B. Improvement in COPD management by access to asthma/COPD clinics in primary care: data from the observational PATHOS study. Respir Med. 2014 Sep;108(9):1345-54. doi: 10.1016/j.rmed.2014.06.002. Epub 2014 Jun 17. PMID 25002194
- [Derived] Janson C, Larsson K, Lisspers KH, Stallberg B, Stratelis G, Goike H, Jorgensen L, Johansson G. Pneumonia and pneumonia related mortality in patients with COPD treated with fixed combinations of inhaled corticosteroid and long acting beta2 agonist: observational matched cohort study (PATHOS). BMJ. 2013 May 29;346:f3306. doi: 10.1136/bmj.f3306. PMID 23719639
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1072&filename=CSP-NIS-RSE-DUM-2010-1.pdf
- See also: CSR-NIS-RSE-DUM-2010-1.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1072&filename=CSP-NIS-RSE-DUM-2010-1.pdf
- See also: NIS-RSE-DUM-2010/1 Clinical Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1072&filename=NCT01146392_CSR_Synopsis_120906.pdf